CLINICAL TRIAL: NCT07244614
Title: Observational Study Assessing the Biosimilar of Ustekinumab in Active Mucocutaneous Behçet's Syndrome Refractory or Intolerant to Conventional Approaches
Brief Title: Ustekinumab in BEhçet's Syndrome STudy
Acronym: USBEST
Status: Recruiting | Type: Observational
Sponsor: Groupe français d'étude des Maladies Inflammatoires de loeil (Other)
Responsible Party: Sponsor
Other Study IDs: USBEST; 2025-A01077-42 (Other: ANSM)
Record Dates: First submitted 2025-09-26; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Behçet's Syndrome (BS)
Keywords: Behçet's syndrome; biosimilar; ustekinumab; refractory; apremilast
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ustekinumab group: patients who have received the Ustekinumab
- Apremilast group: patients who have received the Apremilast

SUMMARY:
This non-interventional study is an observational cohort with parallel groups aiming primarily to describe the success of biosimilar of ustekinumab in Behçet's syndrome in whom conventional approaches have failed or are not suitable well tolerated, and then to compare with patients receiving apremilast within routine care.

Ustekinumab previously prescribed subcutaneously at 90 mg on Week 0, 4, 12 and 20 within the standard of care.

Following non-opposition to participate, patients data will be collected, which will comprise data of the 3-month interval medical visits, except for the first month of treatment, in which the short-term tolerance of treatments is usually assessed (ie, baseline visit, then week 4, 12, 24, 36 and 52). Clinical examination, biological tests and relevant clinical scores (BDCAF, BSAS and PhGA) data that were performed within routine care. No changes to patients' usual care will be made (no additional visits, additional examinations or questionnaires), their safety and well-being remaining therefore unchanged. Data will be collected from the participant's medical record (containing medical reports and examinations, biological tests, nursing records, etc.), for the period of participation in the research, with the only purpose of meeting the objectives of the research. Data will be collected using an electronic 'eCRF observation book on the REDCap platform. The following data will be collected: demographic data (age, sex, weight, height); clinical data (history of the disease, pathology diagnosed, activity of the pathology), treatments, biological data, adverse events. No genetic data will be collected as part of the study. No data will be transferred abroad. No additional questionnaires, examinations or visits will be added by the research. Activity indexes for BS will be calculated as part of routine care. The number, duration and intensity of oral ulcers of patients will be verified by the nurse or the site investigator according to the routine care.

Patients' data with active mucocutaneous Behçet's manifestations with an indication of starting apremilast within standard of care (according to AMM and PNDS) will be retrospectively collected in order to establish a retrospective cohort for comparative purposes.

DETAILED DESCRIPTION:
This non-interventional study is an observational and comparative cohort aiming to describe the success of biosimilar of ustekinumab in Behçet's syndrome in whom conventional approaches have failed or are not suitable well tolerated. Data on 208 patients is expected to be identified as follows:

* data of 104 patients will be collected from patients who have received the ustekinumab
* data of 104 patients will be collected from patients who have received the apremilast.

Ustekinumab is usually prescribed subcutaneously at 90 mg on Week 0, 4, 12 and 20 within the standard of care.

Following non-opposition to participate, patients data will be collected retrospectively according to local clinical practices and usual care, which usually comprises 3-month interval medical visits, except for the first month of treatment, in which the short-term tolerance of treatments is usually assessed (ie, baseline visit, then week 4, 12, 24, 36 and 52). Available data on clinical examination, biological tests and relevant clinical scores (BDCAF, BSAS and PhGA) that are performed within routine care will be retrieved. No changes to patients' usual care will be made (no additional visits, additional examinations or questionnaires), their safety and well-being remaining therefore unchanged. Data will be collected from the participant's medical record (containing medical reports and examinations, biological tests, nursing records, etc.), for the period of participation in the research, with the only purpose of meeting the objectives of the research. Data will be collected using an electronic eCRF observation book on the REDCap platform. The following data will be collected: demographic data (age, sex, weight, height); clinical data (history of the disease, pathology diagnosed, activity of the pathology), treatments, biological data, adverse events. No genetic data will be collected as part of the study. No data will be transferred abroad. No additional questionnaires, examinations or visits will be added by the research. Activity indexes for BS are usually calculated as part of routine care. The number, duration and intensity of oral ulcers of patients might be verified by the nurse or the site investigator according to the routine care.

Patients data with active mucocutaneous Behçet's manifestations with an indication of starting apremilast within standard of care will be also retrospectively collected in order to establish a comparative group, using the same parameters above mentioned

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Non-opposition to study;
* Use of contraceptive measures;
* Fulfillment of the international classification criteria for Behçet's disease, revised in 2013;
* Indication for ustekinumab or apremilast within the standard of care of mucocutaneous Behçet's syndrome
* For ustekinumab cohort: Active mucocutaneous manifestations of Behçet's syndrome that are recurrent, intolerant or refractory to colchicine or apremilast, including oral ulcers, genital ulcers, skin lesions (e.g., pseudofolliculitis), and/or inflammatory arthralgia/arthritis.
* For apremilast cohort: recurrent active mucocutaneous manifestations of Behçet's syndrome naïve of treatment.

Due to its fluctuant characteristics over time, active oral ulcers are defined as two or more oral ulcers over the month preceding inclusion and must have occurred at least three times in the previous 12-month period, despite the previous use of colchicine

Exclusion Criteria:

* Pregnancy;
* Previous treatment failure to ustekinumab;
* Contraindications to ustekinumab, such as:
* Active chronic infections (e.g., active tuberculosis, replicative hepatitis B, HIV, etc.) or malignancies;
* Live vaccins in the past 3 months;
* Severe renal impairment (CrCl <30mL/min/1,73m²)
* Severe hepatic impairment (transaminases 5 times the upper normal values)
* Severe cytopenias:

Platelets < 50 x 103/mm3 Neutrophils < 1000/mm3 Hemoglobin < 8 g/Dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups will be established in this observational cohort:
  1. Patients with active mucocutaneous manifestations of Behçet's syndrome that are either relapsing, refractory or intolerant to conventional treatments, that have received an indication of ustekinumab according to the standard of care of tertiary centres.
  2. Patients with active mucocutaneous manifestations of Behçet's syndrome treated by apremilast within standard of care will be also retrospectively collected in order to establish a comparative group.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Success at Week 24 will be defined as the absence of active mucocutaneous manifestations | Week 24
  Success at Week 24 will be defined as the absence of active mucocutaneous manifestations at week 24 without treatment discontinuation due to inefficacy or toxicity.

SECONDARY OUTCOMES:
Area under the curve (AUC) for the cumulative number of oral ulcers | Week 24
  Area under the curve (AUC) for the cumulative number of oral ulcers along the study period at W24.
Duration (days) of oral and genital ulcers | Week 24
  Duration (days) of oral and genital ulcers up to W24
Number of oral and genital ulcers | Week 24
  Number of oral and genital ulcers up to week 24
Number of painful and swollen joints | Week 24
  Number of painful and swollen joints up to W24
Rate of patients with complete response (ie, no mucocutaneous manifestations), partial response (>50% reduction in overall mucocutaneous manifestations), and no response | Week 12 and Week 24
  Rate of patients with complete response (ie, no mucocutaneous manifestations), partial response (>50% reduction in overall mucocutaneous manifestations), and no response (ie, persistence of mucocutaneous manifestations not fulfilling complete or partial response definitions) at W12 and W24
Rate of treatment discontinuations for safety reasons | Week 24
  Rate of treatment discontinuations for safety reasons up to W24
Rate of treatment failures | Week 24
  Rate of treatment failures (i.e., persistence of active mucocutaneous manifestations that require a change in immunomodulatory therapy) up to W24
Change in BDCAF scores | Week 24
  The score is between 0 and 12. Higher scores indicate a worse evaluation
Frequency and severity of adverse events | 48 months
  Frequency and severity of adverse events (CTCAE grade) along the study period.
Safety of patients receiving the Apremilast | 48 months
  frequency and severity of adverse events in patients receiveing apremilast.
pain intensity (0-10 EVA score) for genital and oral ulcers | WEEK24
  pain intensity (0-10 EVA score) for genital and oral ulcers up to W24
Change in BSAS scores | week24
  The score is between 0 and 100. Higher scores indicate a worse evaluation
Change PhGA scores | week 24
  The score is between 0 and 10. Higher scores indicate a worse evaluation

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU BORDEAUX Hôpital Saint-André - Service de médecine interne, Bordeaux
  - Service de médecine interne-APHP - Henri Mondor, Créteil
  - HOPITAL CROIX-ROUSSE - HCL - service de médecine interne, Lyon
  - Hospices civils de Lyon, Lyon
  - GHSIF Melun, Melun
  - AP-HP-Hôpital COCHIN, Paris
  - service de dermatologie - APHP - St Louis, Paris
  - CHU Rouen_Hôpital Charles Nicolle, Rouen
  - CHU de Rouen - service dermatologie, Rouen
  - APHP_Hopital Lariboisière, Paris, Île-de-France Region
  - APHP_ Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region